CLINICAL TRIAL: NCT06292676
Title: Learning Skills for Emergency Home Delivery
Brief Title: Emergency Home Delivery. Learning Skills for Medical Doctors and Nurses. Kirkpatrick Levels of Learning
Acronym: ERdeliv
Status: Recruiting | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Claudio Celentano, Director, G. d'Annunzio University
Other Study IDs: ObGynEASC004
Record Dates: First submitted 2024-02-26; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Home Birth Delivery
Keywords: home birth; emergency; skills
MeSH Terms: conditions — Emergencies | interventions — Emergency Service, Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: skills retained for home birth delivery in emergency — skills on mannequin for home birth scenario in emergency

SUMMARY:
Mannequin training for emergency home delivery on medical doctors and nurses

DETAILED DESCRIPTION:
two groups will be exposed to frontal lecture and simulato scenario on emergency home birth. After the first training a debriefing will be done. Following a second scenario will bi performed. All participants will complete a google form questionnaire before and after addressed to understand the value of their participation.

ELIGIBILITY:
Inclusion Criteria:

* medical doctors and nurses

Exclusion Criteria:

* none

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: volunteers
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Kirkpatrick levels improvement | 3 months
  improvement knowledge of birth assistance (Kirkpatrick levels value)

CONTACTS AND LOCATIONS:
Locations (1):
- Claudio Celentano, Pescara, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
volunteers undergoing course for emergency home birth
Supporting Information: Study Protocol, ICF
Time Frame: 3 months
Access Criteria: google form